CLINICAL TRIAL: NCT03515707
Title: Autologous Transplant as Treatment for Favorable or Intermediate Risk MRD-Negative AML Patients After Initial Induction Therapy
Brief Title: Stem Cell Transplant to Treat Patients With Favorable or Intermediate Risk Minimal Residual Disease Negative Acute Myeloid Leukemia
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: PI recommended closure
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9784; NCI-2017-02069 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9784 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH); RG9217025 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2018-04-23; First posted 2018-05-03 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Acute Myeloid Leukemia; Minimal Residual Disease Negativity
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Busulfan; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (busulfan, etoposide, ASCT) (Experimental): Patients receive busulfan IV or oral every 6 hours on days -7 to -4 and etoposide IV on day -3. Patients then undergo autologous stem cell transplant on day 0.
  Interventions: Procedure: Autologous Hematopoietic Stem Cell Transplantation; Drug: Busulfan; Drug: Etoposide; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Procedure: Autologous Hematopoietic Stem Cell Transplantation — Undergo ASCT
  Other Names: Autologous Hematopoietic Cell Transplantation; Autologous Stem Cell Transplantation
Drug: Busulfan — Given IV or oral
  Other Names: 1, 4-Bis[methanesulfonoxy]butane; BUS; Bussulfam; Busulfanum; Busulfex; Busulphan; CB 2041; CB-2041; Glyzophrol; GT 41; GT-41; Joacamine; Methanesulfonic Acid Tetramethylene Ester; Methanesulfonic acid, tetramethylene ester; Mielucin; Misulban; Misulfan; Mitosan; Myeleukon; Myeloleukon; Myelosan; Mylecytan; Myleran; Sulfabutin; Tetramethylene Bis(methanesulfonate); Tetramethylene bis[methanesulfonate]; WR-19508
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16-213; VP-16; VP-16-213
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial studies how well autologous stem cell transplant works in treating patients with favorable or intermediate risk, minimal residual disease (MRD)-negative, acute myeloid leukemia. Giving chemotherapy before a peripheral blood stem cell transplant helps kill any cancer cells that are in the body. After treatment, stem cells are collected from the patient's blood and stored. Higher dose chemotherapy is then given to prepare the bone marrow for the stem cell transplant. The stem cells are then returned to the patient to replace the blood-forming cells that were destroyed by the chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the estimated probability of relapse at 2 years after autologous peripheral blood stem cell (PBSC) transplant.

SECONDARY OBJECTIVES:

I. Estimate the probability of transplant-related mortality (TRM) at 100 days following autologous stem cell transplant (ASCT).

II. Estimate probabilities of overall and disease-free survival. III. Assess if biological and molecular correlative studies can predict better outcome.

OUTLINE:

Patients receive targeted busulfan intravenously (IV) or oral (PO) every 6 hours on days -7 to -4 and etoposide IV on day -3. Patients then undergo autologous stem cell transplant on day 0.

After completion of study treatment, patients are followed up yearly for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* AML favorable or intermediate ELN risk
* Achieved true 1st complete response (CR) (absolute neutrophil count [ANC] and platelet count > 1,000/ul and 100,000/ul respectively) after first cycle of induction therapy, with no minimal residual disease (MRD)
* No measurable residual disease (MRD) as assessed by flow cytometry after initial induction therapy
* Performance score Eastern Cooperative Oncology Group (ECOG) 0, 1 or 2
* Creatinine < 2.0 mg/dl and calculated by Cockcroft-Gault (CG) formula or 24 hour measured creatinine clearance (CRCL) > 50
* Not pregnant
* Received 1-2 courses of post remission "consolidation" therapy prior to mobilization PBSC
* No MRD by flow, cytogenetics, fluorescence in situ hybridization (FISH) and molecular testing prior to collection of autologous PBSC collection
* Plan is to collect at least 3 x 10^6 CD34+ PBSC/kg cryopreserved; preference is 4-5 X 10^6 CD34 cells/kg

Exclusion Criteria:

* Life expectancy is severely limited by diseases other than AML
* Total bilirubin > 2.0 mg/dl or serum glutamic-oxaloacetic transaminase (SGOT)/serum glutamate pyruvate transaminase (SGPT) > 2.5 x upper limit of normal (ULN)
* History of Gilbert's disease
* Uncontrolled arrhythmias, left ventricular ejection fraction (LVEF) < 50% or corrected diffusion capacity of the lung for carbon monoxide (DLCO) < 50%
* Significant active infection that precludes transplant
* Hepatitis B or C viremia at time of ASCT
* History of central nervous system (CNS) involvement with AML

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2022-04-15 (Estimated); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
Relapse | Assessed up to 2 years post autologous stem cell transplant (ASCT)
  Proportion of patients who relapse, as defined by 2017 National Comprehensive Cancer Network (NCCN ) Acute Myeloid Leukemia (AML) guidelines.
Treatment related mortality | From first dose of study therapy to day +100
  Number of deaths without a prior relapse (unrelated to disease)

SECONDARY OUTCOMES:
Disease-free survival | Assessed up to 4 years post-ASCT
  Proportion of patients living without relapse
Overall survival | Assessed up to 4 years post-ASCT
  Proportion of patients living with or without relapse

CONTACTS AND LOCATIONS:
Overall Officials: Leona A. Holmberg, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No